CLINICAL TRIAL: NCT04061486
Title: Sperm Separation Efficiency to Maximize Pregnancy Rates: MACS vs. FERTILE Chip
Acronym: FERTIMACS
Status: Completed | Type: Observational
Sponsor: Vida Recoletas Sevilla (Other)
Collaborators: IVI Madrid (Other)
Responsible Party: Sponsor
Other Study IDs: 1904-SEV-050-CR
Record Dates: First submitted 2019-08-16; First posted 2019-08-19 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Infertility, Male
Keywords: MACS; DNA fragmentation; Sperm selection
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental arm: One half of the oocyte cohort is microinjected with sperm selected by the Fertile technique, while the other half of the patient's oocyte cohort is microinjected with sperm selected by the MACS technique.

SUMMARY:
The goal of this observational study is to compare clinical outcomes of two techniques for sperm cell sorting, microfluidic sorting and magnetic activated cell sorting (MACS) technique, in males with high DNA fragmentation within an assisted reproductive treatment. The main questions it aims to answer are:

* Does microfluidic sorting improve pregnancy rate compared to MACS?
* Does microfluidic sorting improve fertilization rate compared to MACS?
* Does microfluidic sorting improve implantation rate compared to MACS?
* Does microfluidic sorting improve blastocyst development rate compared to MACS?

Participants will deposit an eyaculate sample that will be analyzed for DNA fragmentation using a aliquot, then split in two to perform MACS and the microfluidic sorting. Both will be tested for DNA fragmentation (aliquotes) and used for the ICSI treatment with donor oocytes.

Researchers will compare both techniques to see if the selection of the best functional spermatozoa with less DNA fragmentation and clinical outcomes improve.

DETAILED DESCRIPTION:
In assisted reproductive technology (ART), the diagnosis of male infertility has been conducted based on the assessment and analysis of sperm concentration, motility and morphology with the aim of obtaining the best quality of spermatozoa. Any type of damage present in sperm DNA can lead to ART failure. Sperm DNA fragmentation might be the most frequent cause of paternal DNA anomaly transmitted to offspring, and is found in a variable percentage of spermatozoa in subfertile and infertile men. Such DNA fragmentation is negatively correlated with semen quality and consequently, there is a need to develop sperm separation techniques that facilitate retrieval of as many spermatozoa with normal DNA integrity as possible from ejaculated semen.

Because of centrifugation steps associated to swim-up or density-gradient can induce sperm DNA fragmentation via reactive oxygen species (ROS), microfluidic sperm sorters are being used to isolate motile human spermatozoa based on fluid dynamics. It seems to be that using this separation method, spermatozoa do not undergo added physical stress from sources such as a centrifuge. Hence, this new technology has been proposed to minimize DNA damage. In this study, we aim to determine if microfluidic sorting improves the selection of the best functional and with lower DNA fragmentation spermatozoa when compared to magnetic activated cell sorting (MACS) in split semen samples, and increases clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Oocyte recipient patients

Exclusion Criteria:

* Sperm concentration < 5 Mill/ml
* Percentage of motile sperm < 15%

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile patients needing an IVF treatment
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2022-01-09 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | Mar 2019 - Oct 2021
  Total of positive pregnancies / total of patients with embryo transfer

SECONDARY OUTCOMES:
Fertilization rate | Mar 2019 - Oct 2021
  Total of oocyte fertilized / total of oocyte injected
Implantation rate | Mar 2019 - Oct 2021
  Total of implanted embryos / total of transferred embryos
Blastocyst rate | Mar 2019 - Oct 2021
  Total of bastocyst / total of oocyte fertilized

CONTACTS AND LOCATIONS:
Overall Officials: Cristina González Ravina, PhD, Principal Investigator — IVI RMA Seville
Locations (1):
- IVI RMA Seville, Seville, Spain